CLINICAL TRIAL: NCT04871113
Title: A Phase 2a Multicentre, Randomized, Open-Label, Two-Part Adaptive Design Study to Evaluate the Antiviral Effect, Safety and Tolerability of GSK3810109A, an HIV-1 Specific Broadly Neutralizing Human Monoclonal Antibody in Antiretroviral-naïve HIV-1-Infected Adults
Brief Title: A Study to Evaluate the Antiviral Effect, Safety and Tolerability of GSK3810109A in Viremic Human Immunodeficiency Virus (HIV)-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 207959
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: HIV Infections
Keywords: Antiretroviral-naïve; Broadly neutralizing antibody; GSK3810109A; HIV; N6LS
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: The is a sequential treatment, two-part study which will include a screening phase, a randomized monotherapy phase and a standard of care follow-up phase.
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1:GSK3810109A 40milligram(mg)/kilogram intravenously (IV) (Experimental): Participants with human immunodeficiency viruses-1 (HIV-1) received GSK3810109A as a single intravenous (IV) infusion of 40 milligrams per kilogram (mg/kg) dose based on individual bodyweight on Day 1 in part 1.
  Interventions: Biological: GSK3810109A
- Part 1: GSK3810109A 280 mg IV (Experimental): Participants with HIV-1 received GSK3810109A as a single IV infusion of 280 mg dose on Day 1 in part 1.
  Interventions: Biological: GSK3810109A
- Part 2: GSK3810109A 700 mg IV (Experimental): Participants with HIV-1 received GSK3810109A as a single IV infusion of 700 mg dose on Day 1 in part 2. This included dose level determined based on the data of part 1.
  Interventions: Biological: GSK3810109A
- Part 2: GSK3810109A 70 mg IV (Experimental): Participants with HIV-1 received GSK3810109A as a single IV infusion of 70 mg dose on Day 1 in part 2. This included dose level determined based on the data of part 1.
  Interventions: Biological: GSK3810109A
- Part 2: GSK3810109A 700 mg subcutaneously (SC) (Experimental): Participants with HIV-1 received GSK3810109A as a subcutaneous (SC) injection of total 700 mg dose administered as three equally divided SC injections of 2.33 mL each (approximately 7 mL) in quick succession at same time on Day 1 in part 2. This included dose level determined based on the data of part 1.
  Interventions: Biological: GSK3810109A
- Standard of care (SOC) - GSK3810109A 40mg/kg IV (Experimental): Participants who completed the monotherapy phase of treatment of GSK3810109A 40mg/kg IV entered SOC phase to receive dolutegravir + lamivudine regimen as a SOC treatment on SOC Day 1 if deemed appropriate by the investigator and consistent with local guidelines.
  Interventions: Biological: Dolutegravir+lamivudine SOC regimen
- SOC - GSK3810109A 280 mg IV (Experimental): Participants who completed the monotherapy phase of treatment of GSK3810109A 280 mg IV entered SOC phase to receive dolutegravir + lamivudine regimen as a SOC treatment on SOC Day 1 if deemed appropriate by the investigator and consistent with local guidelines.
  Interventions: Biological: Dolutegravir+lamivudine SOC regimen
- SOC - GSK3810109A 700 mg IV (Experimental): Participants who completed the monotherapy phase of treatment of GSK3810109A 700 mg IV entered SOC phase to receive dolutegravir + lamivudine regimen as a SOC treatment on SOC Day 1 if deemed appropriate by the investigator and consistent with local guidelines.
  Interventions: Biological: Dolutegravir+lamivudine SOC regimen
- SOC - GSK3810109A 70 mg IV (Experimental): Participants who completed the monotherapy phase of treatment of GSK3810109A 70 mg IV entered SOC phase to receive dolutegravir + lamivudine regimen as a SOC treatment on SOC Day 1 if deemed appropriate by the investigator and consistent with local guidelines.
  Interventions: Biological: Dolutegravir+lamivudine SOC regimen
- SOC - GSK3810109A 700 mg SC (Experimental): Participants who completed the monotherapy phase of treatment of GSK3810109A 700 mg SC entered SOC phase to receive dolutegravir + lamivudine regimen as a SOC treatment on SOC Day 1 if deemed appropriate by the investigator and consistent with local guidelines.
  Interventions: Biological: Dolutegravir+lamivudine SOC regimen

INTERVENTIONS:
Biological: GSK3810109A — GSK3810109A available as sterile aqueous solution.
  Arms: Part 1: GSK3810109A 280 mg IV; Part 1:GSK3810109A 40milligram(mg)/kilogram intravenously (IV); Part 2: GSK3810109A 70 mg IV; Part 2: GSK3810109A 700 mg IV; Part 2: GSK3810109A 700 mg subcutaneously (SC)
Biological: Dolutegravir+lamivudine SOC regimen — Dolutegravir+lamivudine regimen administered in consistence with investigator input and local guidelines
  Arms: SOC - GSK3810109A 280 mg IV; SOC - GSK3810109A 70 mg IV; SOC - GSK3810109A 700 mg IV; SOC - GSK3810109A 700 mg SC; Standard of care (SOC) - GSK3810109A 40mg/kg IV

SUMMARY:
This study is to evaluate antiviral activity, efficacy, safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of GSK3810109A in HIV-1 infected treatment naive adults. Participants will receive a single dose of GSK3810109A administered either intravenously (IV) or subcutaneously (SC). The study includes a screening phase, a randomized monotherapy phase and a standard of care follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants must have HIV-1 infection within 45 days of the Screening Visit: Plasma HIV-1 RNA greater than or equal to (>=) 5000 copies/mL (c/mL).
* Confirmed screening CD4+ T-cell count >= 350 cells per cubic millimeter (cells/mm3).
* Antiretroviral naïve: No Antiretroviral therapy (ARTs) (in combination or monotherapy) received after the diagnosis of HIV-1 infection.
* Body weight >= 50 kg to less than or equal to (<=) 115 kg.
* Male and/or female. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. All participants participating in the study should be counselled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g. male condom) and on the risk of HIV transmission to an uninfected partner; a. Participants who are female at birth are eligible to participate if at least one of the following conditions applies: Not Pregnant or breastfeeding and at least one of the following conditions applies: Is not a participant of childbearing potential (POCBP). OR Is a POCBP and using an acceptable contraceptive method during the intervention period (at a minimum until after the last dose of study intervention). The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. A POCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) on Day 1, prior to the first dose of study intervention. If a urine test cannot be confirmed as negative (example [e.g.], an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Corrected QT interval (QTc) Interval <= 450 milliseconds (msec)
* Capable of giving signed informed consent.

Exclusion Criteria:

* Participants with primary HIV infection, evidenced by acute retroviral syndrome (e.g., fever, malaise, fatigue, etc) and/or evidence of recent (within 3 months) documented viremia without antibody production and/or evidence of recent (within 3 months) documented seroconversion.
* Participants who are pregnant, breastfeeding, plan to become pregnant or breastfeed during the study.
* The participant has an underlying skin disease or disorder (example i.e. infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria) that would interfere with assessment of injection sites.
* Known history of cirrhosis with or without viral hepatitis co-infection.
* History of clinically relevant hepatitis within last 6 months.
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antigen antibody (anti-HBs) and HBV Deoxyribonucleic acid (DNA) as follows: Participants positive for HBsAg are excluded; Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded. Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and negative for HBV DNA are not excluded.
* Participants with Hepatitis C co-infection.
* Untreated syphilis infection (positive rapid plasma reagin [RPR] at screening) without documentation of treatment. Participants who are one month post completed treatment are eligible if recruitment is open.

Rescreening is allowed after treatment.

* Prior receipt of licensed or investigational monoclonal antibody.
* Any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease except cutaneous Kaposi's sarcoma not requiring systemic therapy.
* Known or suspected moderate or severe hepatic impairment (Class C as determined by Child-Pugh Classification) coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease at the discretion of the investigator.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the study medical monitor for inclusion of the participant prior to randomization.
* Any pre-existing physical or mental condition which, in the opinion of the investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations, or which may compromise the safety of the participant.
* Participants with substance abuse disorders or social restraints that the investigator considers to be possible deterrents to successful completion of the study.
* Participants who in the investigator's judgment, pose a significant suicidality risk. Participants' history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* History of sensitivity to any of the study medications or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Any condition which, in the opinion of the investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs, combination ART or render the participant unable to take oral medication.
* Participants with a positive Corona Virus Disease 2019 (COVID-19) test at Screening. Participants with known COVID-19 positive contacts within the past 14 days, or with symptoms suggestive of active COVID-19 (fever, cough, myalgias, shortness of breath, loss of taste or smell), should be excluded. Participants who remain symptom-free for at least 14 days after a COVID-19 exposure are allowed.
* Has received any HIV-1 immunotherapeutic vaccine or prophylactic vaccine.
* Treatment with any of the following agents within 28 days of screening: radiation therapy; cytotoxic chemotherapeutic agents; any systemic immune suppressant;
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of IP.
* Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.
* Participant enrolled in a prior or concurrent clinical study that includes a drug intervention within the last 30 days.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's inclusion in the study of an investigational compound.
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening period to verify a result.
* ALT >= 3 times the upper limit of normal (ULN).
* Creatinine clearance of <50 mL/minute/1.73 meter^2) via Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) method.
* The participant has a tattoo or other dermatological condition overlying potential injection sites which may interfere with interpretation of injection site reactions or administration of GSK3810109A.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (20):
- United States (6):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Dallas, Texas
- Argentina (5):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Juan
- Brazil (2):
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Canada (4):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
- Mexico (2):
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Monterrey
- GSK Investigational Site, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Derived] Leone PA, Ferro A, Rolle CP, Lupo S, McGowan J, Klein M, Cahn P, Benson P, Griesel R, Warwick-Sanders M, Sanchez M, D'Agostino R, Bettacchi C, Schneider S, Wannamaker P, Dorey D, Wilches V, Gartland M, Brown K, Gandhi Y, Donatti C, Losos J. VH3810109 Efficacy, Safety, Pharmacokinetics, and Incidence of Antidrug Antibodies in Adults With HIV-1 Naive to Antiretroviral Therapy: BANNER Study Results. J Infect Dis. 2025 Dec 20;232(6):e1022-e1032. doi: 10.1093/infdis/jiaf450. PMID 40892985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 unique participants were enrolled in the study including one participant that was re-screened. This re-screened participant signed two different informed consent forms, therefore this participant was counted as enrolling twice.
Pre-assignment Details: Monotherapy phase had 2 parts (Part 1 and 2) where participants received GSK3810109A. All participants who completed monotherapy phase entered standard of care (SOC) follow-up phase to receive a regimen of dolutegravir + lamivudine.
Groups:
- SOC - GSK3810109A 40mg/kg IV: Participants who completed the monotherapy phase of treatment of GSK3810109A 40mg/kg IV entered SOC phase to receive dolutegravir + lamivudine regimen as a SOC treatment on SOC Day 1 if deemed appropriate by the investigator and consistent with local guidelines.
Period: Part1:Monotherapy Phase(up to Day 84)
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC) | SOC - GSK3810109A 40mg/kg IV | SOC - GSK3810109A 280 mg IV | SOC - GSK3810109A 700 mg IV | SOC - GSK3810109A 70 mg IV | SOC - GSK3810109A 700 mg SC
Started (1 participant was randomized to Part 1: GSK3810109A 280 mg IV, but received GSK3810109A 40mg/kg IV intervention. Hence the participant was included in Part 1:GSK3810109A 40milligram(mg)/kilogram intravenously (IV) in the safety and pharmacokinetic set, and in Part 1: GSK3810109A 280 mg IV group in Full ANalysis Set, resulting in different sizes of these populations.) | 8 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 8 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part2:Monotherapy Phase(up to Day 84)
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC) | SOC - GSK3810109A 40mg/kg IV | SOC - GSK3810109A 280 mg IV | SOC - GSK3810109A 700 mg IV | SOC - GSK3810109A 70 mg IV | SOC - GSK3810109A 700 mg SC
Started | 0 | 0 | 16 (Part 2 enrolled new participants and the dosing for part 2 was based on the part 1 data.) | 16 (Part 2 enrolled new participants and the dosing for part 2 was based on the part 1 data.) | 16 (Part 2 enrolled new participants and the dosing for part 2 was based on the part 1 data.) | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 16 | 16 | 16 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SOC Follow-up (SOC Day 1 to 48 Weeks)
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC) | SOC - GSK3810109A 40mg/kg IV | SOC - GSK3810109A 280 mg IV | SOC - GSK3810109A 700 mg IV | SOC - GSK3810109A 70 mg IV | SOC - GSK3810109A 700 mg SC
Started | 0 | 0 | 0 | 0 | 0 | 8 (Participants are transferred from GSK3810109A 40 mg/kg IV arm.) | 6 (Participants are transferred from GSK3810109A 280 mg IV arm.) | 16 (Participants are transferred from GSK3810109A 700 mg IV arm.) | 16 (Participants are transferred from GSK3810109A 70 mg IV arm.) | 16 (Participants are transferred from GSK3810109A 700 mg SC arm.)
Completed | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 14 | 16 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC) | Total
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16 | 62
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 34.3 (9.39) | 34.0 (14.83) | 31.2 (10.46) | 32.3 (10.33) | 31.5 (11.08) | 32.2 (10.62)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 0 | 1 | 4
  Male | 8 | 5 | 14 | 16 | 15 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 1 | 3
  Black or African American | 2 | 1 | 3 | 3 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  White - Arabic/ North African Heritage | 0 | 0 | 0 | 1 | 3 | 4
  White - White/ Caucasian/ European Heritage | 6 | 5 | 10 | 8 | 9 | 38
  Multiple | 0 | 0 | 3 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Decline From Baseline in Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) Levels - Monotherapy Phase
Description: Plasma samples were collected for quantitative analysis of plasma HIV-1 RNA. Maximum decline from baseline in plasma HIV-1 RNA were measured in participants. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. End of Monotherapy Phase is defined as the timepoint when a participant had reached the monotherapy endpoint criteria or a maximum of 84 days follow-up, whichever occurred first.
Time Frame: Baseline (Day 1) and up to Day 84 or end of Monotherapy Phase
Population: The analysis was performed on the safety population, which included all participants who received at least one dose of study treatment. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Copies per milliliter (copies/mL)
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Copies per milliliter (copies/mL)
  Baseline (Day 1) | 12258.5 [1351 to 173710] | 30833.0 [5938 to 104585] | 25466.0 [7180 to 110387] | 25689.5 [7225 to 683576] | 23146.0 [131 to 181078]
  Maximum decline from baseline (up to Day 84/end of Monotherapy Phase): number analyzed (Participants) | 8 | 6 | 15 | 16 | 16
  Maximum decline from baseline (up to Day 84/end of Monotherapy Phase) | -12014.5 [-171577 to -1312] | -26826.5 [-103583 to -5899] | -25966.0 [-107218 to -6944] | -14720.5 [-197793 to -4382] | -12584.0 [-178423 to -69]

2. Primary Outcome: Number of Participants With Adverse Events (AEs) - Monotherapy Phase
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. End of Monotherapy Phase is defined as the timepoint when a participant had reached the monotherapy endpoint criteria or a maximum of 84 days follow-up, whichever occurred first.
Time Frame: Up to Day 84 or end of Monotherapy Phase
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Participants | 7 | 4 | 9 | 8 | 11

3. Primary Outcome: Number of Participants With Worst-case Maximum Grade 2-4 Increase in Post-baseline Values of Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) Compared to the Baseline Values - Monotherapy Phase
Description: Blood samples were collected for the analysis of ALT and AST parameters. The parameters ALT and AST were graded using the Division of Acquired Immunodeficiency Syndrome (DAIDS) criteria Version 2.1 where grades were defined based on numeric criteria as follows Grade 0: participants with missing baseline values; Grade 1: Mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates greater severity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Data of number of participants with 2-4 grade increase at worst-case post-baseline (maximum grade increase post-baseline) is presented. End of Monotherapy Phase is defined as the timepoint when a participant had reached the monotherapy endpoint criteria or a maximum of 84 days follow-up, whichever occurred first.
Time Frame: Baseline (Day 1) and up to Day 84 or end of Monotherapy Phase
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Participants
  ALT, Baseline, Grade 0 | 8 | 6 | 15 | 12 | 15
  ALT, Baseline, Grade 1 | 0 | 0 | 1 | 2 | 1
  ALT, Baseline, Grade 2 | 0 | 0 | 0 | 2 | 0
  ALT, Baseline, Grade 3 | 0 | 0 | 0 | 0 | 0
  ALT, Baseline, Grade 4 | 0 | 0 | 0 | 0 | 0
  ALT, Worst Case Post-Baseline, Increase to Grades 2 to 4 | 0 | 0 | 0 | 0 | 0
  ALT, Worst Case Post-Baseline, Increase to Grades 3 to 4 | 0 | 0 | 0 | 0 | 0
  AST, Baseline, Grade 0 | 8 | 6 | 15 | 14 | 16
  AST, Baseline, Grade 1 | 0 | 0 | 0 | 1 | 0
  AST, Baseline, Grade 2 | 0 | 0 | 1 | 1 | 0
  AST, Baseline, Grade 3 | 0 | 0 | 0 | 0 | 0
  AST, Baseline, Grade 4 | 0 | 0 | 0 | 0 | 0
  AST, Worst Case Post-Baseline, Increase to Grades 2 to 4 | 1 | 0 | 1 | 0 | 1
  AST, Worst Case Post-Baseline, Increase to Grades 3 to 4 | 1 | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Treatment-emergent Abnormal Electrocardiogram (ECG) Findings - Monotherapy Phase
Description: A 12-lead ECG were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QT interval corrected using Fridericia's formula (QTcF) intervals. ECG findings were categorized as normal, abnormal clinically significant (CS) and abnormal not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of participants with abnormal (CS and NCS) ECG findings are presented. End of Monotherapy Phase is defined as the timepoint when a participant had reached the monotherapy endpoint criteria or a maximum of 84 days follow-up, whichever occurred first.
Time Frame: Up to Day 84 or end of Monotherapy Phase
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Participants
  Abnormal - Clinically Significant | 0 | 0 | 0 | 0 | 0
  Abnormal - Not Clinically Significant | 3 | 2 | 3 | 4 | 7

5. Primary Outcome: Number of Participants With Grade 2-4 Injection Site Reactions (ISR) - Monotherapy Phase
Description: Number of participants with grade 2-4 injection site reactions are presented. The ISR were graded using the Division of Acquired immunodeficiency syndrome (DAIDS) criteria Version 2.1 where grades were defined based on numeric criteria as follows Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates more severe condition. End of Monotherapy Phase is defined as the timepoint when a participant had reached the monotherapy endpoint criteria or a maximum of 84 days follow-up, whichever occurred first.
Time Frame: Up to Day 84 or end of Monotherapy Phase
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Day 14 (AUC [0-14]) of GSK3810109A - Monotherapy Phase
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3810109A.
Time Frame: Pre-dose (Day 1), 3 and 24 hours post-dose on day 1, days 3, 6, 9, 11, and 14
Population: Analysis was performed on the Pharmacokinetic (PK) population, which included all participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values with the actual dose and PK sampling time will be considered as non-missing values).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day *microgram/millilitre (day*ug/mL)
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 14 | 16 | 16
Day *microgram/millilitre (day*ug/mL) | 5346.3194 (29.6508) | 690.8944 (53.2785) | 1181.1688 (24.4990) | 212.6213 (79.1478) | 493.0579 (55.0909)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK3810109A - Monotherapy Phase
Description: Cmax is defined as maximum observed concentration of GSK3810109A.
Time Frame: Pre-dose (Day 1), 3 and 24 hours post-dose on day 1, days 3, 6, 9, 11, and 14
Population: Analysis was performed on the PK population, which included all participants in the Safety population who had at least 1 non-missing PK assessment (NQ values with the actual dose and PK sampling time will be considered as non-missing values).
Measure: Mean (Standard Deviation); unit: Microgram/millilitre (μg/mL)
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Microgram/millilitre (μg/mL) | 1131.5000 (329.91168) | 131.1500 (86.65425) | 243.0625 (57.37301) | 42.7688 (54.32691) | 45.0938 (20.48930)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of GSK3810109A - Monotherapy Phase
Description: Tmax is defined as time to reach Cmax
Time Frame: Pre-dose (Day 1), 3 and 24 hours post-dose on day 1, days 3, 6, 9, 11, and 14
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Days | 0.0385 [0.024 to 0.125] | 0.1233 [0.026 to 0.149] | 0.0340 [0.021 to 0.128] | 0.0278 [0.003 to 0.994] | 5.9177 [1.884 to 14.966]

9. Secondary Outcome: Plasma Concentration at Day 14 (C14) of GSK3810109A - Monotherapy Phase
Description: Blood samples were collected at indicated time point for pharmacokinetic analysis of GSK3810109A.
Time Frame: At Day 14
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 11 | 11 | 15
μg/mL | 221.45 (23.76) | 27.49 (49.24) | 55.30 (22.08) | 7.98 (89.70) | 29.52 (54.30)

10. Secondary Outcome: Change From Baseline in Log10 Plasma HIV-1 RNA Relative to Cmax - Monotherapy Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. Statistical analysis for relationship between PK parameter (Cmax) and PD measure (change from baseline in logarithm to base 10 (log10) values for plasma HIV-1 RNA) were explored using an Emax non-linear model. The model parameters estimated included: maximum response (Emax), PK parameter value that attains 50 percent (%) of the maximal effect (EC50) and residual variability (s2e). End of Monotherapy Phase is defined as the timepoint when a participant had reached the monotherapy endpoint criteria or a maximum of 84 days follow-up, whichever occurred first.
Time Frame: Baseline (Day 1) and up to Day 84 or end of Monotherapy Phase
Population: The analysis was performed on the safety population, which included all participants who received at least one dose of study treatment. Only those participants with data available at the specified time points were analyzed. Only participants in the IV dosing group with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter (copies/mL)
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV
Number analyzed (Participants) | 8 | 6 | 16 | 16
Log10 copies per milliliter (copies/mL)
  Baseline (Day 1) | 4.139 (0.6433) | 4.493 (0.4800) | 4.465 (0.3594) | 4.582 (0.6144)
  Change from baseline (up to Day 84 or end of Monotherapy Phase) | 0.091 (0.2359) | -0.357 (0.4191) | -0.110 (0.1940) | -0.179 (0.4319)
Statistical Analysis 1: Comparison: Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) vs Part 1: GSK3810109A 280 mg IV vs Part 2: GSK3810109A 700 mg IV vs Part 2: GSK3810109A 70 mg IV; Test type: Other; Emax = -1.848, 95% CI 2-sided [-2.225 to -1.472] — Emax is defined as maximum response
Statistical Analysis 2: Comparison: Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) vs Part 1: GSK3810109A 280 mg IV vs Part 2: GSK3810109A 700 mg IV vs Part 2: GSK3810109A 70 mg IV; Test type: Other; EC50 = 68.578, 95% CI 2-sided [15.866 to 121.290] — EC50 is defined as the dose (in mg) that attains the 50% of the maximal effect
Statistical Analysis 3: Comparison: Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) vs Part 1: GSK3810109A 280 mg IV vs Part 2: GSK3810109A 700 mg IV vs Part 2: GSK3810109A 70 mg IV; Test type: Other; s2e = 0.257, 95% CI 2-sided [0.145 to 0.368] — e is defined as random error assumed to be normally distributed with mean zero and constant variance (s2)

11. Secondary Outcome: Absolute Values of Cluster of Differentiation 4 Plus (CD4+) and CD8+ T Cell Counts - Monotherapy Phase
Description: Blood samples were collected as prespecified. CD4+ and CD8+ T cell counts were assessed using flow cytometry. End of Monotherapy Phase is defined as the timepoint when a participant had reached the monotherapy endpoint criteria or a maximum of 84 days follow-up, whichever occurred first.
Time Frame: From Day 1 (Baseline) and up to Day 84 or end of Monotherapy Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cells per cubic milimeter
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Cells per cubic milimeter
  CD4+, Baseline (Day 1 (Monotherapy Phase) | 360.5 (166.54) | 412.8 (120.85) | 427.3 (187.22) | 467.3 (194.45) | 476.7 (180.28)
  CD4+, Day 84/end of Monotherapy Phase | 392.3 (196.16) | 443.0 (155.17) | 424.0 (171.33) | 412.9 (98.50) | 462.4 (276.72)
  CD8+, Baseline (Day 1 (Monotherapy Phase) | 852.0 (441.83) | 884.5 (389.42) | 781.8 (303.75) | 1161.3 (697.24) | 898.0 (348.48)
  CD8+, Day 84/End of Monotherapy Phase | 837.9 (482.68) | 869.8 (376.86) | 744.0 (267.73) | 993.1 (394.84) | 765.9 (296.18)

12. Secondary Outcome: Absolute Values of CD4+ and CD8+ T Cell Counts - SOC Phase
Description: Blood samples were collected as prespecified. CD4+ and CD8+ T cell counts were assessed using flow cytometry.
Time Frame: Up to Week 48 (SOC Phase)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cells per cubic milimeter
Arm/Group | SOC - GSK3810109A 40mg/kg IV | SOC - GSK3810109A 280 mg IV | SOC - GSK3810109A 700 mg IV | SOC - GSK3810109A 70 mg IV | SOC - GSK3810109A 700 mg SC
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Cells per cubic milimeter
  CD4+, Week 48 (SOC Phase) | 500.5 (211.17) | 601.0 (44.74) | 580.9 (165.29) | 671.3 (180.25) | 723.9 (300.24)
  CD8+, Week 48 (SOC Phase) | 685.9 (308.89) | 738.4 (213.22) | 684.9 (286.60) | 856.0 (325.04) | 816.6 (364.40)

13. Secondary Outcome: Change From Baseline in CD4+ and CD8+ T Cell Counts - Monotherapy Phase
Description: as for outcome 11
Time Frame: Up to Day 84 or end of Monotherapy Phase (compared with baseline [Day 1])
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cells per cubic milimeter
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Cells per cubic milimeter
  CD4+, Baseline (Day 1 (Monotherapy Phase) | 360.5 (166.54) | 412.8 (120.85) | 427.3 (187.22) | 467.3 (194.45) | 476.7 (180.28)
  CD4+, Day 84/end of Monotherapy Phase (compared with baseline): number analyzed (Participants) | 8 | 6 | 16 | 16 | 15
  CD4+, Day 84/end of Monotherapy Phase (compared with baseline) | 31.8 (48.27) | 30.2 (79.83) | -3.3 (125.78) | -54.3 (121.18) | -19.6 (166.64)
  CD8+, Baseline (Day 1 (Monotherapy Phase) | 852.0 (441.83) | 884.5 (389.42) | 781.8 (303.75) | 1161.3 (697.24) | 898.0 (348.48)
  CD8+, Day 84/end of Monotherapy Phase (compared with baseline): number analyzed (Participants) | 8 | 6 | 16 | 16 | 15
  CD8+, Day 84/end of Monotherapy Phase (compared with baseline) | -14.1 (213.24) | -14.7 (281.75) | -37.8 (206.05) | -168.2 (401.82) | -105.7 (246.85)

14. Secondary Outcome: Change From Baseline in CD4+ and CD8+ T Cell Counts - SOC Phase
Description: Blood samples were collected as prespecified. CD4+ and CD8+ T cell counts were assessed using flow cytometry.
Time Frame: Up to Week 48 (SOC Phase)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cells per cubic milimeter
Arm/Group | SOC - GSK3810109A 40mg/kg IV | SOC - GSK3810109A 280 mg IV | SOC - GSK3810109A 700 mg IV | SOC - GSK3810109A 70 mg IV | SOC - GSK3810109A 700 mg SC
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Cells per cubic milimeter
  CD4+, Baseline (Day 1 (Monotherapy Phase) | 360.5 (166.54) | 412.8 (120.85) | 427.3 (187.22) | 467.3 (194.45) | 476.7 (180.28)
  CD4+, Week 48 of SOC Phase (compared with baseline): number analyzed (Participants) | 8 | 5 | 14 | 14 | 16
  CD4+, Week 48 of SOC Phase (compared with baseline) | 140.0 (91.08) | 180.4 (114.37) | 134.9 (205.13) | 233.8 (174.02) | 247.3 (230.95)
  CD8+, Baseline (Day 1 (Monotherapy Phase) | 852.0 (441.83) | 884.5 (389.42) | 781.8 (303.75) | 1161.3 (697.24) | 898.0 (348.48)
  CD8+, Week 48 of SOC Phase (compared with baseline): number analyzed (Participants) | 8 | 5 | 14 | 14 | 16
  CD8+, Week 48 of SOC Phase (compared with baseline) | -166.1 (274.92) | -159.4 (275.37) | -119.7 (198.49) | -217.5 (490.10) | -81.4 (230.95)

15. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) Against GSK3810109A - Monotherapy Phase
Description: Serum samples were collected to analyze the presence of ADAs against GSK3810109A using validated immunoassays. End of Monotherapy Phase is defined as the timepoint when a participant had reached the monotherapy endpoint criteria or a maximum of 84 days follow-up, whichever occurred first.
Time Frame: At Day 1 and Day 84 or end of Monotherapy Phase
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 8 | 6 | 16 | 16 | 16
Participants
  Baseline (Day 1): number analyzed (Participants) | 8 | 6 | 15 | 16 | 16
  Baseline (Day 1) | 0 | 0 | 0 | 0 | 0
  Day 84/End of Monotherapy Phase: number analyzed (Participants) | 8 | 5 | 16 | 16 | 16
  Day 84/End of Monotherapy Phase | 1 | 2 | 0 | 3 | 0

16. Secondary Outcome: Number of Participants With Positive ADAs Against GSK3810109A - SOC Phase
Description: Serum samples were collected to analyze the presence of ADAs against GSK3810109A using validated immunoassays.
Time Frame: At Week 48 (SOC Phase)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SOC - GSK3810109A 40mg/kg IV | SOC - GSK3810109A 280 mg IV | SOC - GSK3810109A 700 mg IV | SOC - GSK3810109A 70 mg IV | SOC - GSK3810109A 700 mg SC
Number analyzed (Participants) | 8 | 5 | 14 | 16 | 16
Participants | 0 | 0 | 1 | 2 | 0

17. Secondary Outcome: Titers of Positive ADAs Against GSK3810109A - Monotherapy Phase
Description: as for outcome 15
Time Frame: At Day 84 or end of Monotherapy Phase
Population: as for outcome 1
Measure: Median (Full Range); unit: Titers
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC)
Number analyzed (Participants) | 1 | 2 | 0 | 3 | 0
Titers | 40 [40 to 40] | 60 [40 to 80] |  | 80 [40 to 640] |

18. Secondary Outcome: Titers of Positive ADAs Against GSK3810109A - SOC Phase
Description: Serum samples were collected to analyze the presence of ADAs against GSK3810109A using validated immunoassays.
Time Frame: At Week 48 (SOC Phase)
Population: as for outcome 1
Measure: Median (Full Range); unit: Titers
Arm/Group | SOC - GSK3810109A 40mg/kg IV | SOC - GSK3810109A 280 mg IV | SOC - GSK3810109A 700 mg IV | SOC - GSK3810109A 70 mg IV | SOC - GSK3810109A 700 mg SC
Number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
Titers |  |  | 40 [40 to 40] | 160 [160 to 160] |

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 12 weeks for Monotherapy Phase (Part 1 and Part 2 groups) and up to 48 weeks for SOC Phase (SOC groups).
Description: Safety population included all participants who received at least one dose of study treatment.
Arm/Group | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) | Part 1: GSK3810109A 280 mg IV | Part 2: GSK3810109A 700 mg IV | Part 2: GSK3810109A 70 mg IV | Part 2: GSK3810109A 700 mg Subcutaneously (SC) | SOC - GSK3810109A 40mg/kg IV | SOC - GSK3810109A 280 mg IV | SOC - GSK3810109A 700 mg IV | SOC - GSK3810109A 70 mg IV | SOC - GSK3810109A 700 mg SC
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/16 | 0/16 | 0/16 | 0/8 | 0/6 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/16 | 0/16 | 0/16 | 1/8 | 0/6 | 3/16 | 2/16 | 4/16
Other Adverse Events (participants affected / at risk) | 7/8 | 4/6 | 9/16 | 8/16 | 11/16 | 8/8 | 3/6 | 12/16 | 13/16 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) (N=8) | Part 1: GSK3810109A 280 mg IV (N=6) | Part 2: GSK3810109A 700 mg IV (N=16) | Part 2: GSK3810109A 70 mg IV (N=16) | Part 2: GSK3810109A 700 mg Subcutaneously (SC) (N=16) | SOC - GSK3810109A 40mg/kg IV (N=8) | SOC - GSK3810109A 280 mg IV (N=6) | SOC - GSK3810109A 700 mg IV (N=16) | SOC - GSK3810109A 70 mg IV (N=16) | SOC - GSK3810109A 700 mg SC (N=16)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Human rhinovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1:GSK3810109A 40milligram(mg)/Kilogram Intravenously (IV) (N=8) | Part 1: GSK3810109A 280 mg IV (N=6) | Part 2: GSK3810109A 700 mg IV (N=16) | Part 2: GSK3810109A 70 mg IV (N=16) | Part 2: GSK3810109A 700 mg Subcutaneously (SC) (N=16) | SOC - GSK3810109A 40mg/kg IV (N=8) | SOC - GSK3810109A 280 mg IV (N=6) | SOC - GSK3810109A 700 mg IV (N=16) | SOC - GSK3810109A 70 mg IV (N=16) | SOC - GSK3810109A 700 mg SC (N=16)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Application site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal human papilloma virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monkeypox (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proctitis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Viral sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helminthic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilloma viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Secondary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myokymia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chemical burn of gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal ulcer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT04871113/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT04871113/SAP_001.pdf